CLINICAL TRIAL: NCT02317172
Title: Efficacy of Novel Edible Gel-based Artificial Saliva in Thai Geriatric Populations With Systemic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dental Innovation Foundation Under Royal Patronage (Other)
Collaborators: Thammasat University (Other); Srinakharinwirot University (Other); Mahidol University (Other); Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DIF-03
Record Dates: First submitted 2014-12-11; First posted 2014-12-15 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Xerostomia; Hypertension; Diabetes Mellitus
Keywords: Saliva substitute; Edible gel; Xerostomia; Diabetes Mellitus; Hypertension
MeSH Terms: conditions — Xerostomia; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gel-based artificial saliva (Experimental): Continuous oral intake of edible gel-based artificial saliva (30-50 ml/day) for four weeks
  Interventions: Other: Gel-based artificial saliva

INTERVENTIONS:
Other: Gel-based artificial saliva — Gel-based artificial saliva is a novel gel-like, edible moisturizing gel designed to relieve dry mouth.
  Other Names: Oral moisturizing jelly

SUMMARY:
Elderly people usually have systemic diseases and take medications that can cause dry mouth. The purpose of this study is to determine whether continuous use of edible, gel-based artificial saliva in geriatric population with dry mouth problems will reduce signs and symptoms of dry mouth and improve quality of patients' saliva.

DETAILED DESCRIPTION:
A pre-post test trial was conducted in 120 elders with xerostomia. All subjects received a total of 50 ml (10ml x 5 times) OMJ per day. Subjective and objective dry mouth scores, salivary pH, buffering capacity and satisfaction were monitored at 2 weeks and 1 month use, compared to baseline. The data were analyzed by Repeated Measure ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Have systemic diseases such as hypertension or diabetes mellitus and take medications that can cause dry mouth
* Report symptoms of dry mouth

Exclusion Criteria:

* Subjects with uncontrolled systemic diseases
* Subjects who aspirate upon eating
* Subjects who smoke
* Subjects who are allergic to component of the intervention

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Changes in subjective dry mouth score | baseline, 2 weeks and 4 weeks after intervention
  The outcome measure (subjective dry mouth score) will be measured before and 2 and 4 weeks after continuous usage of edible gel-based artificial saliva (30-50 ml/day for at least 5 days per week)

SECONDARY OUTCOMES:
Changes in objective dry mouth score | baseline, 2 weeks and 4 weeks after intervention
  The outcome measure will be measured before and 2 and 4 weeks after continuous usage of edible gel-based artificial saliva (30-50 ml/day for at least 5 days per week)
Changes in salivary Potential of Hydrogen ion (pH) | baseline, 2 weeks and 4 weeks after intervention
  The outcome measure will be measured before and 2 and 4 weeks after continuous usage of edible gel-based artificial saliva (30-50 ml/day for at least 5 days per week)
Changes in salivary buffering capacity | baseline, 2 weeks and 4 weeks after intervention
  The outcome measure will be measured before and 2 and 4 weeks after continuous usage of edible gel-based artificial saliva (30-50 ml/day for at least 5 days per week)
Satisfaction of the edible gel-based artificial saliva | at the first day of trial
  All subjects will try a few spoon of the edible gel based saliva and a commercially available inedible gel-based saliva. Then, all subjects will be interviewed for satisfaction of both products and compare the results.

CONTACTS AND LOCATIONS:
Overall Officials: Aroonwan Lam-ubol, DDS, PhD, Principal Investigator — Srinakharinwirot University
Locations (1):
- Department of Health, Ministry of Health, Nonthaburi, Thailand

REFERENCES:
- [Derived] Dalodom S, Lam-Ubol A, Jeanmaneechotechai S, Takamfoo L, Intachai W, Duangchada K, Hongsachum B, Kanjanatiwat P, Vacharotayangul P, Trachootham D. Influence of oral moisturizing jelly as a saliva substitute for the relief of xerostomia in elderly patients with hypertension and diabetes mellitus. Geriatr Nurs. 2016 Mar-Apr;37(2):101-9. doi: 10.1016/j.gerinurse.2015.10.014. Epub 2015 Nov 26. PMID 26631691